CLINICAL TRIAL: NCT04121182
Title: Prevention of pneumonIA in Nursing hOme
Acronym: PIANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/17/0452
Record Dates: First submitted 2019-08-19; First posted 2019-10-09 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Pneumonia
Keywords: Nursing home; Prevention
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Seven thousand residents will be recruited by 280 nursing home in 2 major regions in France and followed for 1 year. At the end of the randomization, half of the institutions will benefit from an "on-line" training on the prevention and management of pulmonary disease in residents. Other institutions will continue their usual practice (routine care) and will not benefit from training during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing home with On-line training (Experimental): 25 randomized residents will be included by nursing home Half of the institutions (randomized too) will benefit from an "on-line" training on the prevention and management of resident lung diseases
  Interventions: Other: On-line training
- Nursing home with usual practice (Active Comparator): This group of Institutions continue their usual practice (routine care) and will not benefit from training during the study period.
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: On-line training — Nursing teams randomized in the intervention group will benefit from an intervention in the form of a specific training "online" on the prevention of pneumonia and their management in the nursing home This training focuses on prevention, and management during the infectious period (the false food route and the management of pneumonia).
  Arms: Nursing home with On-line training
Other: Usual practice — Nursing home with usual practice : The act of comparison is defined by the usual care, as they are performed in the nursing home at the time of the study. No restrictions are placed on residents or caregivers of any kind in the care of the resident.
  Arms: Nursing home with usual practice

SUMMARY:
Infections in nursing home are associated with high morbidity and mortality. Pulmonary infections are known to be the most problematic. In our INCUR observational study of 773 residents, 20.13% of residents had pneumonia during the year of follow-up. On average, the extra cost of pneumopathies was 4,467 euros / patient for the long-term care facility and 3,044 euros for the hospital.

DETAILED DESCRIPTION:
The pneumopathies in nursing home are the main cause of hospitalization of residents. Depending on the series, 9 to 50% of residents with pneumonia should be transferred. This reflects the difficulties faced by nursing home care teams in these situations. The respiratory symptomatology of nursing home residents is difficult to grasp and the prescribed antibiotic therapy is often considered inappropriate (25% to 75% of cases). Prevention of resident pneumonia, such as vaccination against pneumococcus remains poorly practiced, influenza vaccination teams or vitamin D supplementation.

In addition to the risk of mortality, lung diseases are often the cause of a rapid functional decline. Preventing pneumonia in nursing homes is therefore an important issue in the prevention of dependence, the quality of life, the health care system (use of hospitalization and transfer to emergencies) and health expenditure. In this vulnerable population, a prevention intervention seems particularly relevant.

In this research project, the investigators hypothesize that a multi-domain prevention intervention for pneumonia carried out by nursing teams in nursing homes can reduce the incidence of pneumonia. They also believe that this action would reduce emergency transfers and health expenditures.

ELIGIBILITY:
Inclusion Criteria:

* Living in a nursing home for at least 30 days at the start of inclusions,
* Having received information concerning the study and having not expressed opposition to participate,
* For which an agreement in principle of the attending physician has been obtained.

Exclusion Criteria:

* Refusal of the resident (or of his legal representative) or of his treating physician after given information,
* Resident at the end of life (life expectancy evaluated within one month by the coordinating physician),
* Resident whose attending physician is already involved in the PIANO study under a resident of another nursing home.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3818 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
The comparison of the incidence of lung disease number between the two groups | 1 year
  After the one-year : to compare of the incidence of lung disease between the two groups of Nursing home (the on-line formation/casual care) The diagnosis of pneumopathy will be defined on the criteria of the Infectious Risk Observatory in Geriatrics that are appropriate for nursing home residents, with at least two of the criteria defined for pneumonia
Number of Medical evidence of rattles or crepitates | 1 year
  Medical evidence of rattles or crepitates on chest auscultation : rattles or crepitates are criteria for the diagnosis of pneumopathy

SECONDARY OUTCOMES:
Establish a differential cost-effectiveness ratio at 1 year of the care of the residents in nursing home | 1 year
  Establish a differential cost-effectiveness ratio at 1 year of the care of the residents in nursing home by a healthcare team trained in the management of pneumonia in the context of E-learning training versus usual care.
  The medico-economic analysis will consist in a cost-effectiveness evaluation of a training in the prevention of pneumopathies aimed at the carers in nursing homes, compared to the usual practice.
Evaluation of the time spent by the health care team to support the patient between two groups | 1 year
  Perform an evaluation of the time spent by the health care team to support the patient for Basic Activities of Daily Living (ADL), Instrumental Activities of Daily Living, supervision of care and patient monitoring. They will use the Questionnaire adapted from Resource Utilization in Dementia - Formal Care (RUD-FOCA)
Evaluating the incidence of all-cause hospitalizations | 1 year
  Evaluating the incidence of number of all-cause hospitalizations to compare with the hospitalizations due to pneumonia
Evaluate the evolution of quality of care indicators in the nursing home | 1 year
  Indicators of quality of care in the nursing home related to the risk of pneumonia will be reported at T-2 months and T12 months. These indicators will be provided by the coordinating physician :
  * Vaccination rate (Residents; Staff).
  * Presence in the nursing home of a protocol for taking care of the false route
  * In case of pneumopathy, the use of antibiotic therapy will be indicated
Functional decline of residents | 1year
  The degree of dependence of the residents will be evaluated by the carers of the nursing home by the Scale ADL (Basic Activity Daily Living) of Katz during 12 months On this scale of 0 (totally dependent) to 6 points (independent), a difference of 0.5 points would be considered clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Rolland, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France